CLINICAL TRIAL: NCT00110110
Title: Multicenter Phase II Study for International Intraocular Retinoblastoma Classification Groups B, C & D Tumors Treated With Carboplatin-Etoposide-Vincristine-Cyclosporine-Focal Therapy Multimodality Protocol (OCRN Multicenter RB 2003)
Brief Title: Combination Chemotherapy and Cyclosporine Followed by Focal Therapy for Bilateral Retinoblastoma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Collaborators: Terry Fox Foundation (Other)
Responsible Party: Principal Investigator, Helen Chan, Oncologist, The Hospital for Sick Children
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1000005587; HFSC-OCRN-RB-2003 (Other: The Hospital for Sick Children); CDR0000422340 (Other: The Hospital for Sick Children)
Record Dates: First submitted 2005-05-03; First posted 2005-05-04 (Estimated); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Retinoblastoma
Keywords: intraocular retinoblastoma
MeSH Terms: conditions — Retinoblastoma | interventions — Filgrastim; Granulocyte Colony-Stimulating Factor; Carboplatin; Cyclosporine; Etoposide; Vincristine; Cryosurgery; Cryotherapy; Laser Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- CEV Chemo + Cyclosporine & Focal Therapy (Experimental): Systemic carboplatin (28 mg/kg/dose), etoposide (12 mg/kg/dose) and vincristine sulfate (0.025 mg/kg/dose for the first cycle and 0.05 mg/kg/dose for subsequent cycles if first cycle well-tolerated) chemotherapy given with cyclosporin A (33 mg/kg/dose). Following 4-6 cycles CEV chemotherapy (depending on tumor stage) given every 3 weeks, focal laser therapy and/or cryosurgery are applied for tumor consolidation. Filgrastim is given after each chemotherapy cycle to prevent severe neutropenia.
  Interventions: Biological: filgrastim; Drug: Carboplatin; Drug: Cyclosporine; Drug: Etoposide; Drug: vincristine sulfate; Procedure: cryosurgery; Procedure: laser therapy

INTERVENTIONS:
Biological: filgrastim — Given after chemo cycle for 7 days or until neutrophil counts return to normal.
  Other Names: granulocyte colony-stimulating factor (G-CSF)
Drug: Carboplatin — Given at 28 mg/kg/dose.
Drug: Cyclosporine — Given at 33 mg/kg/dose
Drug: Etoposide — Given at 12 mg/kg/dose
Drug: vincristine sulfate — Given at 0.025 mg/kg/dose for the first cycle and 0.05 mg/kg/dose for subsequent cycles if first cycle well-tolerated
  Other Names: vincristine
Procedure: cryosurgery — Local application of extreme cold to destroy residual tumor.
  Other Names: cryotherapy
Procedure: laser therapy — Local and precise application of laser beams to destroy residual tumor.

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as carboplatin, etoposide, and vincristine, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Sometimes when chemotherapy is given, it does not stop the growth of tumor cells. The tumor is said to be resistant to chemotherapy. Giving cyclosporine together with chemotherapy may reduce drug resistance and allow the tumor cells to be killed. Cryotherapy kills tumor cells by freezing them. Laser therapy uses light to kill tumor cells. Giving combination chemotherapy together with cyclosporine followed by cryotherapy and/or laser therapy may be an effective treatment for retinoblastoma.

PURPOSE: This phase II trial is studying how well giving combination chemotherapy together with cyclosporine followed by cryotherapy and/or laser therapy works in treating patients with newly diagnosed retinoblastoma in both eyes.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare the efficacy of neoadjuvant high-dose carboplatin and etoposide, vincristine, and cyclosporine (CSA) followed by ophthalmic focal therapy comprising cryotherapy and/or laser therapy to historical world data of chemotherapy treatment without CSA, in terms of increasing the proportion of eyes that remain relapse free and do not require external beam radiotherapy and/or enucleation, in patients with newly diagnosed Group B, C, or D bilateral intraocular retinoblastoma.

Secondary

* Determine the toxicity of this regimen in these patients.

OUTLINE: This is a multicenter study.

Patients receive high-dose carboplatin IV over 30 minutes on day 1; vincristine IV over 5 minutes and high-dose etoposide IV over 25 minutes on day 2; cyclosporine IV over 1 hour before chemotherapy and then over 2 hours after chemotherapy on days 1 and 2, and filgrastim (G-CSF) subcutaneously once daily beginning on day 3 and continuing until day 16 or until blood counts recover. Treatment repeats every 21 days for a total of 3 courses for patients with Group B disease and a total of 6 courses for patients with Group C or D disease.

Patients undergo eye examination under anesthesia (EUA) at initial staging and then before each course of chemotherapy. Patients with small peripheral tumors in eyes without retinal detachment undergo minimal focal therapy (mainly cryotherapy) during EUA at initial staging and then after chemotherapy courses 1 and 2. At EUA after the third and subsequent courses of chemotherapy, patients with tumors that have sufficiently reduced in size undergo additional cryotherapy or laser therapy. After completion of chemotherapy, patients with any suspicious, active, or reactivated tumor undergo additional cryotherapy and/or laser therapy during EUA approximately every 4-8 weeks (or at longer intervals) for up to 5 years (as needed).

After completion of study chemotherapy, patients are followed every 3 months for 2 years, every 6 months for 2 years, and then annually for 1 year.

PROJECTED ACCRUAL: A total of 71 patients will be accrued for this study within 2.4 years.

ELIGIBILITY:
>>INCLUSION CRITERIA<<

DISEASE CHARACTERISTICS:

* Clinical diagnosis of bilateral intraocular retinoblastoma (RB)

  * International Intraocular Retinoblastoma Classification (IIRC) Group B, C, or D disease in 1 or both eyes
  * IIRC Group E disease in 1 eye allowed provided the eye was enucleated at diagnosis AND there is no extraocular RB in the enucleated eye by histologic confirmation AND there is IIRC Group B, C, or D disease in the remaining eye

PATIENT CHARACTERISTICS:

Age

* Over 30 days

Performance status

* Not specified

Life expectancy

* Not specified

Hematopoietic

* Not specified

Hepatic

* AST and ALT < 2 times upper limit of normal (ULN)
* Conjugated and unconjugated bilirubin < 2 times ULN

Renal

* Creatinine < 1.5 times ULN
* Glomerular filtration rate (GFR) ≥ 100 mL/min* NOTE: *A 4-hour IV hydration is allowed if GFR is low due to poor hydration or transient dehydration

Other

* Meets 1 of the following auditory criteria:

  * Normal audiogram
  * At least normal responses to speech by audiogram
  * Documentation of hearing by acoustic emission test
  * Recording of evoked potentials by auditory brain stem response

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* Not specified

Endocrine therapy

* Not specified

Radiotherapy

* Not specified

Surgery

* See Disease Characteristics

  >>EXCLUSION CRITERIA<<
* IIRC Group A disease in 1 or both eyes
* unilateral RB
* extraocular or metastatic RB
* younger than 30 days
* Glomerular filtration rate (GFR) < 100 mL/min

Min Age: 30 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 71 (Estimated)
Dates: Start 2004-06 (Actual); Primary Completion 2016-04-20 (Actual); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Comparing efficacy of study treatment with historic world data, in terms of increasing the proportion of eyes that remains relapse-free while avoiding external beam radiation and/or enucleation | 5 year follow-up per patient
  Efficacy

SECONDARY OUTCOMES:
Toxicity during treatment | 5 year follow-up per patient
  Toxicity

CONTACTS AND LOCATIONS:
Overall Officials: Brenda L Gallie, MD, Principal Investigator — The Hospital for Sick Children; Elise Heon, MD, Principal Investigator — The Hospital for Sick Children; Helen SL Chan, MD, BS, Study Chair — The Hospital for Sick Children
Locations (6):
- Canada (3):
  - Children's and Women's Hospital of British Columbia, Vancouver, British Columbia
  - Hospital for Sick Children, Toronto, Ontario
  - Montreal Children's Hospital at McGill University Health Center, Montreal, Quebec
- Hospital San Juan de Dios, Santiago, Chile
- Sankara Nethralaya Super Specialty Clinic, Chennai, India
- Kandang Kerbau Women's and Children's Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No